CLINICAL TRIAL: NCT02052115
Title: Behavioral Weight Loss and Exercise After Treatment (BEAT): Predictors of Weight Loss Success in Overweight Breast Cancer Survivors
Brief Title: Behavioral Weight Loss and Exercise After Treatment (BEAT)
Acronym: BEAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kim Dittus, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VCC 1311; 1P20GM103644-01A1 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; exercise; weight loss; executive function; breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise and weight loss (Other): 12 month exercise and weight loss intervention
  Interventions: Behavioral: 12 month exercise and weight loss intervention

INTERVENTIONS:
Behavioral: 12 month exercise and weight loss intervention

SUMMARY:
Overweight and physically inactive breast cancer survivors are at increased risk of breast cancer recurrence and mortality. Cancer treatment-related changes that likely mediate weight loss and exercise success include the long term effects such as fatigue, psychological distress and impaired executive (cognitive) function.

This study will explore the variability in how breast cancer survivors respond to a behavioral weight loss intervention. The primary objectives include determining the degree to which success with a behavioral weight loss intervention in overweight breast cancer survivors is explained by measures of executive function as measured with task performance at 6 and 12 months and associated brain function imaging (fMRI), collected at baseline only.Additionally, the study is designed to determine the degree to which selected measures of cancer-related symptoms account for variance in the success of breast cancer survivors at 6 and 12 months following entry into a behavioral weight loss and exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis
* Received surgery +/- chemotherapy +/- radiation for treatment of a Stage I, II or III breast cancer. Ongoing treatment with monoclonal antibodies and/or anti-estrogen therapy is acceptable
* Completion of initial therapy 6 weeks prior to study initiation
* BMI of 27-45 kg/m^2

Exclusion Criteria:

* Prior diagnosis of malignancy other than non-melanoma skin cancer (i.e. prior non-melanoma skin cancer is not an exclusion criteria)
* Medical conditions that limit food choices such as celiac sprue or inflammatory bowel disease
* Inability to walk on flat ground (or a treadmill) at 2.5 mph for 5 minutes
* Age <21 and >70
* Presence of body metal
* Psychotic or central nervous system impairment that would limit compliance with study requirements, including dementia
* Evidence of metastatic disease
* Symptomatic heart disease (chest pain or equivalent with activity)
* Exercise limiting pulmonary disease or need for oxygen to exercise
* Individuals taking mood stabilizing medications including: Lithium, valproic acid, also called divalproex sodium (Depakote), carbamazepine (Tegretol), lamotrigine (Lamictal), oxcarbazepine (Trileptal), olanzapine (Zyprexa), aripiprazole (Abilify), risperidone (Risperdal), ziprasidone (Geodon), clozapine (clorazil)
* Participants with an active neurologic disorder that affects the central nervous system, including seizures, and Parkinson's disease
* Weight loss of >10 lbs in the previous 6 months
* Participation in > 150 minutes of moderate intensity activity by self report, unless activity level by accelerometer is less than 150 minutes of moderate intensity activity

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of executive function and weight loss success | 12 months
  Determine the degree to which success with a behavioral weight loss intervention in overweight breast cancer survivors is explained by measures of executive function, measured with task performance and associated brain function imaging (fMRI), at 6 and 12 months.

SECONDARY OUTCOMES:
Correlation of cancer related symptoms and weight loss | 12 months
  Determine the degree to which selected measures of cancer-related symptoms account for variance in the success of breast cancer survivors at 6 and 12 months
Efficacy of a weight loss intervention | 12 months
  Determine the effectiveness of a behavioral weight loss and exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dittus, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- Vermont Cancer Center, Burlington, Vermont, United States